CLINICAL TRIAL: NCT04953000
Title: Local, Multicenter, Non-interventional, Ambispective Study in Severe Hemophilia A Patients on Standard and PK-tailored Prophylaxis With Octocog Alfa (Advate®) in the Russian Federation
Brief Title: A Study of Standard and Individualized Prophylactic Treatment With Advate in Men and Boys With Severe Hemophilia A
Acronym: HAPKIDO
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-761-4001; MACS-2020-051901 (Other: Takeda)
Record Dates: First submitted 2021-07-06; First posted 2021-07-07 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants: Male participants with severe or moderate hemophilia A who have been treated with FVIII concentrate octocog alfa (Advate) during at least 12 months prior to the study enrollment, who started octocog alfa treatment in 2021 or currently being treated with octocog alfa will be observed in this study.

SUMMARY:
The main aim of this study is to learn about changes in the lowest blood levels of Factor VIII in men and boys when upgraded from standard prophylaxis with Advate to individualized prophylaxis with Advate.

No study medicines will be provided to participants in this study. The study sponsor will not be involved in how participants are treated but will provide instructions on how the clinics will record what happens during the study. Participants will need to visit the study doctor 3 times in total during the study. During these visits, study data will be collected by the study doctor.

DETAILED DESCRIPTION:
Local, Multicenter, Non-interventional, Ambispective Study in Severe Hemophilia A Patients on Standard and PK-tailored Prophylaxis With Octocog Alfa (Advate®) in the Russian Federation

ELIGIBILITY:
Inclusion Criteria:

* Male participants of all ages with severe hemophilia A (FVIII ˂1%) or moderate hemophilia A with severe bleeding phenotype who:

  * had been on standard prophylaxis or PK-tailored prophylaxis with octocog alfa during at least 12 months prior to the study enrollment (150 participants) or who started Advate® treatment in 2021 (20 participants),
  * is being treated with octocog alfa at the moment of enrolment with any of the above mentioned treatment modalities, and
  * had been assigned octocog alfa provision in Federal reimbursement program 2021
* Availability of participants' records sufficient for data collection according to the study objectives during the retrospective period of the study for participants who had been on standard prophylaxis or PK-tailored prophylaxis with octocog alfa during at least 12 months prior to the study enrollment
* Written informed consent provided by the participant or, in case of children below 14 years of age, by participant's parent or participant's legally acceptable representative.

Exclusion Criteria:

* Failure to obtain the participant's written informed consent
* Participation in any interventional study of products for hemophilia or other hemostasis disturbances treatment during 12 months prior to the study enrollment for participants who has retrospective data collection period and during 12 months after the study enrollment for all participants.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male participants of all ages being treated with octocog alfa (Advate) for severe hemophilia A in 2021 will be enrolled in this study.
Sampling Method: Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2021-08-19 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Time per Week Spent With Factor VIII (FVIII) Trough Level Below 1 Percent (%) on the Standard Prophylaxis and After Pharmacokinetic (PK) -tailored Prophylaxis | From 12 months prior to study enrollment up to Visit 3 (Month 12)
  PK-tailoring prophylaxis is defined as FVIII replacement prophylactic therapy based on PK parameters of each particular participant. Time per week spent with Through FVIII level below 1% on standard and PK-tailored prophylaxis will be reported.

SECONDARY OUTCOMES:
Percentage of Participants With More Than 19 Hours per Week Spent With FVIII Trough Level Below 1% on Standard Prophylaxis Versus on PK-tailored Prophylaxis | From 12 months prior to study enrollment up to Visit 3 (Month 12)
  Percentage of participants with more than 19 hours per week with FVIII trough level below 1% on standard and PK-tailored prophylaxis will be reported.
Percentage of Participants With Upgraded Dosing Regimen Based on PK-assessment | Baseline up to Visit 3 (Month 12)
  Upgraded dosing regimen includes dose upgrade, dosing intervals modification, and/or FVIII trough level upgrade to above 1%. Percentage of participants with upgraded dosing regimen based on PK-assessment will be reported.
Percentage of Time per Week Spent With FVIII Trough Level Below 1%, 1 to less than (<) 3%, and Greater Than or Equal to (>=) 3% While on Standard and Individualized Prophylaxis | From 12 months prior to study enrollment up to Visit 3 (Month 12)
  Individualized prophylaxis is defined as prophylactic therapy based on PK parameters of each individual participant. Percentage of time per week spent with FVIII through level below 1%, 1- <3%, and >=3% while on standard and individualized prophylaxis will be reported.
Percentage of Participants With FVIII Trough Level Permanently Above 1% on Standard Prophylaxis vs on PK-tailored Prophylaxis | From 12 months prior to study enrollment up to Visit 3 (Month 12)
  Percentage of participants with FVIII trough level permanently above 1% on standard and PK-tailored prophylaxis will be reported.
Correlation Between the Time per Week Spent With FVIII Trough Level Below 1% and Spontaneous Annualized Bleeding Rate (ABR) on Standard Prophylaxis | From 12 months prior to study enrollment up to Visit 3 (Month 12)
  Correlation between the time per week spent with FVIII trough level below 1% and spontaneous ABR on standard prophylaxis will be assessed using Pearson's correlation coefficient.
Correlation Between the Time per Week Spent With FVIII Trough Level Below 1% and Spontaneous Annualized Joint Bleeding Rate (AJBR) on Standard Prophylaxis | From 12 months prior to study enrollment up to Visit 3 (Month 12)
  Correlation between the time per week spent with FVIII trough level below 1% and spontaneous AJBR on standard prophylaxis will be assessed using Pearson's correlation coefficient.
Total Consumption of FVIII Before and After PK-tailored Prophylaxis in Participants With Upgraded Dosing Regimen | From 12 months prior to study enrollment up to Visit 3 (Month 12)
  Total consumption of FVIII before and after PK-tailored prophylaxis in participants with upgraded dosing regimen will be reported.
Percentage of Participants With Positive Dynamics of Body Status After Transfer From Standard to Individualized Prophylaxis | Baseline up to Visit 3 (Month 12)
  Positive dynamics of body status is related with increased physical activity (change in body mass index [BMI], waist: hip ratio [WHR]. Percentage of participants with positive dynamics of body status after transfer from standard to individualized prophylaxis will be reported.
Percentage of Participants Categorized Based on Number of Hospitalizations due to Insufficient Bleeding Control Before and After PK-tailored Prophylaxis | From 12 months prior to study enrollment up to Visit 3 (Month 12)
  Percentage of participants categorized based on number of hospitalization due to insufficient bleeding control before and after PK-tailored Prophylaxis will be reported.
Percentage of Participants Categorized Based on Number of Days Away From Work and School/Institute Due to Insufficient Bleeding Control Before and After PK-tailored Prophylaxis | From 12 months prior to study enrollment up to Visit 3 (Month 12)
  Percentage of participants categorized based on number of days away from work and school/institute due to insufficient bleeding control before and after PK-tailored prophylaxis will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (13):
- Russia (13):
  - City Children's Hospital No. 1, Kazan', Tatarstan Republic
  - Chelyabinsk Regional Children's Clinical Hospital, Chelyabinsk
  - Children's Regional Clinical Hospital, Khabarovsk
  - Krasnoyarsk Regional Clinical Center for Maternal and Child Health, Krasnoyarsk
  - Morozovskaya Children's City Clinical Hospital of the Department of Healthcare of the city of Moscow, Moscow
  - State Budgetary Institution of Healthcare "Republican children's clinical hospital" of the Ministry of Health of the Kabardino-Balkar Republic, Nal'chik
  - State Novosibirsk Regional Clinical Hospital, Novosibirsk
  - Regional Children's Clinical Hospital, Rostov-on-Don
  - City Polyclinic No. 37, Saint Petersburg
  - Regional Children's Clinical Hospital No. 1, Vladivostok
  - Volgograd Regional Clinical Oncological Dispensary, Volgograd
  - Voronezh Regional Children's Clinical Hospital No. 1, Voronezh
  - State Autonomous Healthcare Institution of the Sverdlovsk Region "Regional Children's Clinical Hospital", Yekaterinburg

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/60e84d641f1122001e30a94c